CLINICAL TRIAL: NCT05217368
Title: the Effect of Mandala Studies on Fear of Birth Outcomes in Primiparous Pregnant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 886
Record Dates: First submitted 2022-01-21; First posted 2022-02-01 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Fear of Childbirth
Keywords: Mandala; Pregnancy; Primiparous; Antenatal Education
MeSH Terms: interventions — Prenatal Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group/mandala painting (Experimental): Mandala painting will be done in addition to routine antenatal education.
  Interventions: Other: mandala painting; Other: antenatal education
- antenatal education class (No Intervention): Only routine antenatal education will be done.

INTERVENTIONS:
Other: mandala painting — In addition to routine antenatal education, pregnant women included in the experimental group will be asked to practice at least 1 mandala per day at least 5 times a week during the 6-week pregnancy education under the supervision of a researcher.
  Arms: experimental group/mandala painting
Other: antenatal education — Routine antenatal education will be given.
  Arms: experimental group/mandala painting

SUMMARY:
Fear experienced at the time of birth and after birth is considered as fear of childbirth. If the fear occurred before pregnancy or if the pregnancy increases the severity of the fear, this can lead to "Tocophobia". When the literature is examined; In addition to birth preparation education, different methods such as cognitive behavioral theory, analytical theory, psychodrama, haptotherapy and art therapy groups have been found to be effective in reducing fear of birth. No study has been found in the literature on the effect of mandala on fear of birth and birth outcomes. By reducing the women's fear of childbirth of this study; It is predicted that it will reduce the need for medical intervention at birth, increase the normal birth rate, have a more positive birth experience and contribute to the well-being of postpartum women.

DETAILED DESCRIPTION:
This research was planned as a randomized controlled study to determine the effect of mandala studies on fear of labor and delivery results in primiparous pregnant women. We will work with pregnant women who accept to participate in the study among the pregnant women who applied to the online birth and baby preparation training program at the Istanbul Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital Pregnancy Training Center. Since this research was planned experimentally, a power analysis was applied considering the number of pregnant women who applied to the pregnant school of the hospital where the research was conducted in 2020 in order to determine the number of people to be included in each group.( Akın et al. 2018) Sample size, 80% power, 0.05 margin of error, When calculated using the G*Power (3.0.10) Program with an effect level of 0.5, it was determined that at least 48 pregnant women should be recruited for each of the experimental and control groups. Considering that there may be a loss of participants during the study process, it is planned to include 75 pregnant women in both groups, and a total of 150 pregnant women are planned to be included in the study. Randomization of the experimental (n=75) and control (n=75) groups will be provided by the research randomizer.org program.In the study, an introductory information form and Wijma Birth Expectation/Experience (W-DEQ A) scale will be given to the pregnant women who applied to the birth and baby preparation training program to determine the level of fear of birth. Pregnant women with a score of 38 or more will be informed about the subject and invited to the study. During the interview, address and contact information will be obtained from the participants in order to be able to communicate. The forms required for the follow-up of the pregnant women included in the experimental and control groups will be sent to the addresses of the participants by courier in printed form and they will be asked to send them back. In addition to the routine pregnant training, the pregnant women included in the experimental group, at least 5 times a week during the 6 weeks of pregnancy training under the supervision of researcher Tuğba Topcu. They will be asked to do at least 1 mandala work per day. The same mandala study box will be given to each pregnant woman in order to ensure standardization in the pregnant women included in the experimental group. At the end of the training, the researcher Tuğba Topcu will apply the Wijma Birth Expectation/Experience scale to the experimental and control groups in order to determine the level of fear of birth. Postpartum Follow-up Form will be used at the end of delivery, Wijma Birth Expectation/Experience Scale (W DEQ) and Birth Experience Scale will be used to determine the level of birth fear experienced by pregnant women.

Statistical analysis Statistical analysis of the data will be done by using the Statistical Package for the Social Sciences (SPSS) package program and consulting a statistics expert. Apart from the individual characteristics of the individuals included in the study, whether the Wijma Birth Expectation/Experience Scale-Version A, Postpartum Follow-up Chart, Wijma Birth Expectation/Experience Scale-B Version and Birth Experience Scale total scores show a normal distribution; Shapiro Wilks test will be used, if it is found to be normally distributed, mean ± standard deviation will be given as descriptive statistics, and if it is not normally distributed, median (median) and width between quarters values will be given. In the comparison of individual characteristics and scale scores, Independent Sample T test will be applied in independent groups in those with normal distribution, Mann-Whitney U test in independent groups that do not show normal distribution, Paired-Sample T test in dependent groups with normal distribution, and Wilcoxon test in dependent groups that do not show normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Those who want to participate in the study voluntarily,
* Able to speak and understand Turkish,
* Living with his wife,
* Over 18 years old,
* Primiparous pregnant women
* Without a diagnosis of risky pregnancy and,
* Between 24-32 weeks of pregnancy,
* A score of 38 or more on the Wijma Birth Experience/Expectation Scale A,
* Hearing in order to follow group work,
* Those who do not have comprehension and vision problems will be included in the research.

Exclusion Criteria:

* Absence from the 6-week pregnant school for more than one week,
* Less than 30 mandala exercises over 6 weeks those who do,
* Filling in the survey forms incompletely,
* Those who develop any health problems during pregnancy will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy/ Experience Questionnaire Version A (W-DEQ-A) | 6 monts
  It was developed to measure the fear of childbirth. Turkish validity and reliability were done. The scale consists of 33 items. In this scale, there are questions about labor pains and how the birth will be, how they will feel, the feelings when the baby is born, and thoughts about the birth within a month. The answers in the scale are in six-point Likert type numbered from 0 to 5. 0 is evaluated as "totally" and 5 as "not at all". The lowest score obtained from the scale is 0 and the highest score is 165. Wijma Delivery Expectancy/ Experience Questionnaire Version A scores are evaluated over four subgroups. These; Those with low level of fear of childbirth (Wijma-A score ≤ 37), those with moderate fear of childbirth (Wijma-A score between 38-65), those with severe fear of childbirth (Wijma- A scale score 66-84), and those with a clinical degree of fear of childbirth living (Wijma-A scale score ≥ 85).
Wijma Birth Expectation/Experience Scale (W-DEQ) version B: | It is recommended to be administered at least 2 hours after birth and within 15 days at the latest.
  It was developed to measure the fear of childbirth. The scale consists of 32 items. The answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. 0 means "totally" and 5 as "not at all". While the minimum score on the scale is 0, the maximum score is 160. As the score increases, the fear of childbirth experienced by women increases. Questions 2, 3, 6, 7, 10, 11, 14, 18, 19, 23, 24, 26, 30 are calculated by turning them in the opposite direction. The scale, which was adapted into Turkish and validated and reliable, has six sub-dimensions.
Birth Experience Scale | within 1-2 days after delivery
  It is a scale specific to the birth experience, developed for screening purposes and improving the psychological dimension of birth. Birth Experience Scale assesses parents' perceptions of stress, pain, control, fear, and support during childbirth. It is recommended that this evaluation be done in the hospital within 1-2 days immediately after birth. Higher scores indicate a more negative birth experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Topcu T, Bingol FB. Mandala as a New Intervention for Reducing Fear of Childbirth: A Randomized Controlled Trial. J Midwifery Womens Health. 2025 May-Jun;70(3):414-421. doi: 10.1111/jmwh.13722. Epub 2024 Dec 11. PMID 39663544